CLINICAL TRIAL: NCT05678699
Title: The Effects of Medicaid Policy Interventions on Racial Equity in Severe Maternal Morbidity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dara Mendez, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY22080184; 1R01NR020670-01 (NIH)
Record Dates: First submitted 2022-10-26; First posted 2023-01-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Severe Maternal Morbidity; Maternal Death
MeSH Terms: conditions — Maternal Death | interventions — Doulas; Standard of Care

STUDY DESIGN:
Intervention Model Description: Evaluation of policy interventions at the state level comparing within state and across states over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) Only (Other): The investigators will employ a quasi-experimental study design to test two hypotheses: H1: SMM rates among Black people will decline after the interventions (equity payment and obstetric bundled payment), relative to people of other race groups within Pennsylvania (PA); and H2: Racial inequities in SMM will decline among those exposed to the interventions in PA, relative to those in similar states. The investigators will collect qualitative data to assess the effects of the Medicaid healthcare interventions on beneficiaries' experiences.
  Interventions: Behavioral: Medicaid healthcare quality interventions (equity payment and obstetric bundled payment); Behavioral: Standard Care
- Doula Only (Other): The investigators will test two hypotheses: H1: SMM rates among Black people will decline more after the addition of doula care in PA, relative to healthcare quality interventions alone. H2: Racial inequities in SMM will decline more among those exposed to both healthcare quality and doula care interventions in PA, relative to states implementing doula care only. The investigators will collect qualitative data to assess the effects of the Medicaid healthcare and service interventions on beneficiaries' experiences.
  Interventions: Behavioral: Doula; Behavioral: Standard Care
- Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) + Doula (Other)
  Interventions: Behavioral: Medicaid healthcare quality interventions (equity payment and obstetric bundled payment); Behavioral: Doula; Behavioral: Standard Care
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) — This study has two components, with the first component being examined in Aim 1 and the first and second components being examine in aim 2.
  1) health equity incentive payment program makes available $26 million annually in Medicaid managed care organization (MCO) payments to plans that improve access to timely prenatal care and well-child visits among Black beneficiaries. The equity-focused obstetric care bundled payment model provides incentives for clinicians to improve on a wide range of pregnancy health outcomes, and specifically incentivizes improvements among Black beneficiaries
  Arms: Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) + Doula; Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) Only
Behavioral: Doula — This study has two components, with the first component being examined in Aim 1 and the first and second components being examine in aim 2.
  1. health equity incentive payment program makes available $26 million annually in Medicaid managed care organization (MCO) payments to plans that improve access to timely prenatal care and well-child visits among Black beneficiaries. The equity-focused obstetric care bundled payment model provides incentives for clinicians to improve on a wide range of pregnancy health outcomes, and specifically incentivizes improvements among Black beneficiaries.
  2. care intervention by coverage of doula services for all Medicaid beneficiaries across Pennsylvania.
  Arms: Doula Only; Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) + Doula
Behavioral: Standard Care — Participants receive standard care without quality interventions or doula care
  Arms: Doula Only; Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) + Doula; Medicaid healthcare quality interventions (equity payment and obstetric bundled payment) Only

SUMMARY:
The goal of this study is to learn about the effects of structural inventions, such as equity-focused Medicaid polices, on severe maternal morbidity (SMM) and mortality and maternal health. The main questions it aims to answer are:

1. What is the effect of Medicaid healthcare quality interventions on SMM?
2. What is the effect of Medicaid healthcare quality interventions + doula care?
3. What are Medicaid beneficiaries' experiences in receiving services and the potential impact of integration of doula services and equity practices?

Participants will be asked to describe experiences as a result of structural interventions and focused Medicaid policies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and postpartum Medicaid beneficiaries across the US

Qualitative:

* Medicaid beneficiaries who self-identify as Black and/or live in PA Health Equity Zones
* Doulas who provide care to Medicaid beneficiaries in Pennsylvania
* Medicaid Managed Care Organization (MCO) administrators in Pennsylvania. Severe maternal morbidity and mortality outcomes will be assessed in healthcare records and for these quantitative outcomes, patients will not be recruited individually

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000000 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Severe maternal morbidity (SMM) | 20 weeks gestation through 42 days postpartum
  SMM rate based on the Centers for Disease Control algorithm

SECONDARY OUTCOMES:
All cause mortality | Delivery date through one year after delivery
  Binary indicator of mortality based on Social Security Administration records
Follow up for chronic conditions | 43 days through 1 year after delivery
  Percent of persons who receive guideline concordant care for depression, substance use disorders, immunizations, and screening and referral for social determinants of health
Provision of evidence care in pregnancy and postpartum | During pregnancy and postpartum up to 1 year
  Percent of Medicaid patients among each provider who receive screening and follow up for depression, treatment for substance use disorders, perinatal immunizations, and screening and referral for social determinants of health
Medicaid managed care administrator perspectives on policy interventions | Year 3
  Qualitative self report of perspectives

OTHER OUTCOMES:
Assess the changes in effects of the Medicaid healthcare quality interventions on beneficiaries' experiences | Years 2, 3, and 4
  The investigators will collect qualitative data from three different study populations across Pennsylvania who will be affected by the Medicaid policies under study: 1) Medicaid beneficiaries (n=100; Years 2 and 4); 2) Doula care providers (n=60; Years 2 and 4); Managed Care Organization (MCO) leadership (n=10); Year 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh School of Public Health, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No